CLINICAL TRIAL: NCT02763748
Title: the Prospective, Randomized and Comparative Clinical Study of Laparoscopic and Endoscopic Cooperative Surgery in the Treatment of Gastrointestinal Stromal Tumor
Brief Title: the Laparoscopic and Endoscopic Cooperative Surgery of Gastrointestinal Stromal Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-019
Record Dates: First submitted 2016-04-26; First posted 2016-05-05 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Laparoscopic surgery (Experimental): Laparoscopic endoscopy combined surgery. This is a kind of traditional surgical method.
  Interventions: Procedure: Laparoscopic endoscopy combined surgery
- laparoscopic and endoscopic (Experimental): LECS resects the tumor completely by laparoscopy with the help of the precise positioning and guidance of endoscopy .
  Interventions: Procedure: laparoscopic and endoscopic cooperative surgery
- Single-arch laparoscopic and endoscopic (Experimental): Single-arch LECS resects the tumor completely by laparoscopy with the help of the precise positioning and guidance of endoscopy
  Interventions: Procedure: Single-arch laparoscopic and endoscopic cooperative surgery

INTERVENTIONS:
Procedure: Laparoscopic endoscopy combined surgery
  Arms: Laparoscopic surgery
Procedure: laparoscopic and endoscopic cooperative surgery
  Arms: laparoscopic and endoscopic
Procedure: Single-arch laparoscopic and endoscopic cooperative surgery
  Arms: Single-arch laparoscopic and endoscopic

SUMMARY:
Gastric stromal tumor is a gastrointestinal mesenchymal tumor with malignant differentiation potential, the incidence increased year by year. The surgical resection is the primary treatment for it. Although laparoscopic GIST resection has many benefits，due to in lack of the delicate sense of touch, it could lead to the incomplete resection and disorders of digestion. More than 33% of postoperative patients have the gastric dysfunction. Laparoscopic endoscopy combined surgery is different from the past technology. It is a new radical resection of GIST presented by Japanese scholars. LECS resects the tumor completely by laparoscopy with the help of the precise positioning and guidance of endoscopy .This method conforms to the idea of the modern minimally invasive surgery, and avoids many problems，such as incomplete resection and disorders of digestion caused by excessive tissue resection. our team will spearhead the GIST treatment of LECS. First of all, the investigators will collect 120 cases of GIST patients, randomly assigned for the laparoscopic group, the LECS, single-arch the LECS surgical treatment. Secondly, to analyzing the basic treatment and follow-up data, including the operation time, blood loss, the number of transfer laparotomy, the number of cut edge positive, the distances of cut edge away from the tumor edge, the cases of anastomotic fistula bleeding, stenosis, average such confinement, the meal time, cost of treatment, tumor recurrence rate, the presence of residual stomach, upset stomach and frequency, reflux esophagitis, bile reflux gastritis and other indicators.The purpose of this subject is to observe the effectivity and safety of LECS and single-arch the LECS, invent serval LECS equipment patents and provide some references for LECS applying to the minimally invasive surgery of the digestive tract tumor and multidisciplinary treatment mode .

ELIGIBILITY:
Inclusion Criteria:

* Patients without contraindications gastroscope，surgery and anesthesia;
* Gastroscope found submucosal lesions, qualitative hard;Endoscopic ultrasonography (EUS) confirmed the lesions come from the muscularis propria
* Tumors diameter > 2 cm;Or tumors had < 2 cm, but the position is located in the stomach wall, after nearly cardia and it is a difficult position for gastroscope ;
* Tumors diameter < 5 cm, the tumors had complete, no broken feed and bleeding
* Not found the tumor metastasis
* There is no history of abdominal surgery, no severe abdominal cavity adhesion
* Patients signed informed consent

Exclusion Criteria:

* Patients with preoperative assessment of distant metastasis;
* Patients with preoperative radiation and chemotherapy or hormone therapy;
* Patients with acute obstruction, bleeding or perforation of the emergency surgery
* Patients with a history of abdominal trauma or abdominal surgery.
* Patients with contraindications gastroscope，surgery and anesthesia;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence rate | 2 years

SECONDARY OUTCOMES:
the operation time | one hour-five hours
the all number of postoperative complications（ frequency,reflux esophagitis and bile reflux gastritis） | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jun She, M.D.; PhD., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes